CLINICAL TRIAL: NCT03233490
Title: CPR Training in Students to Increase Bystander Intervention in Out-of-hospital Cardiac Arrest.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Leif Svensson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013/358-31
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Coping Skills
Keywords: CPR training; students; willingness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPR training and web corse intervention (Experimental): The students performed a web course (Help Brain Heart) prior training
  Interventions: Other: CPR training
- CPR training intervention (Experimental): CPR training without web course
  Interventions: Other: web course

INTERVENTIONS:
Other: web course — Web course Help Brain Heart was conducted Before CPR training.
  Arms: CPR training intervention
Other: CPR training — No web course was conducted
  Arms: CPR training and web corse intervention

SUMMARY:
The overall aim of this thesis is to identify the factors that may affect 13 year old students' acquisition of CPR skills and their willingness to act. The primary hypothesis is that the training method (intervention) influences the participants' acquisition of practical CPR skills and willingness to intervene.

The study used a cluster randomized design, based on a randomization list generated by an independent statistician. The school classes were randomly assigned to different CPR training interventions.

A strategic sample, where invitation to participate in the study was sent to the headmasters of all council schools, with seventh grade students, in two Swedish municipalities (140,000). Thus, the sample consists of participants with different cultural as well as socio-economic background. Eighteen of 24 schools agreed to participate. Four schools did not respond and two schools had a routine to offer CPR education only for grade nine (all six schools from the same municipality). The eighteen schools who agreed to participate consisted of sixty-eight classes with 1547 students.

Prior to study participation, students and their guardians obtained a letter with study information. Study participation of the individual students was voluntary and all participants gave an oral informed consent.

Inclusion criteria: seventh grade student in one of the participating schools. Exclusion criteria: student does not want to participate, student with a physical handicap that limited the physical performance, classes of students with development disabilities (these classes are age-integrated and have fewer students per class).

DETAILED DESCRIPTION:
The main interventions were app or DVD-based education. In addition to the main intervention some classes were randomized to various additional interventions; web-course, visits of elite athletes, practical test, reflection and AED training. All CPR education was performed in accordance with the ERC guidelines of 2010. Training was given to the entire class together. The classes consisted of 14-29 students. All participants in all intervention groups used an individual training manikin, MiniAnne, during the training. The schools were allowed to keep the training manikins after the end of study. Ten teachers were previous CPR instructors and another 19 teachers received a five hours education to become CPR instructor. All teachers obtained individual oral and written instructions about each class randomized intervention method and written bullet points about how the course would be implemented, to ensure that they were up to date with present guidelines and training. The teachers acted as facilitators; they introduced the lesson, gave advice on the fly, answered questions and completed the course.

ELIGIBILITY:
Inclusion Criteria:

* seventh grade student in one of the participating schools

Exclusion Criteria:

* student does not want to participate
* student with a physical handicap that significantly limited the physical performance
* classes of students with development disabilities (these classes are age integrated and have fewer students per class).

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1547 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2014-10-22 (Actual); Study Completion 2014-10-22 (Actual)

PRIMARY OUTCOMES:
The total score of the modified Cardiff test at six months | At six months follow-up test
  The total score was calculated by adding the individual scores of the 12 different categories (check responsiveness by talking, check responsiveness by shaking, open the airway, checks respiration, dials 112, compression/ventilation ratio, hand-position during compression, average compression depth, total compression counted, average ventilation volume, total ventilation counted, total hands-off time) assessed by the practical test.

SECONDARY OUTCOMES:
The total score of the modified Cardiff test directly after training | Directly after training (on the day of intervention)
  The total score was calculated by adding the individual scores of the 12 different categories (check responsiveness by talking, check responsiveness by shaking, open the airway, checks respiration, dials 112, compression/ventilation ratio, hand-position during compression, average compression depth, total compression counted, average ventilation volume, total ventilation counted, total hands-off time) assessed by the practical test.
Self-reported willingness to make a lifesaving intervention | Both directly after training (on the day of intervention) and at six months
  Self-reported willingness to make a lifesaving intervention was measured by a questionnaire
Knowledge about stroke, acute myocardial infarction and living habits | Both directly after training (on the day of intervention) and at six months
  Theoretical knowledge about acute myocardial infarction and living habits was measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: L Svensson, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No
No data shall be analyzed at the individual level.

REFERENCES:
- [Derived] Hollenberg J, Claesson A, Ringh M, Nordberg P, Hasselqvist-Ax I, Nord A. Effects of native language on CPR skills and willingness to intervene in out-of-hospital cardiac arrest after film-based basic life support training: a subgroup analysis of a randomised trial. BMJ Open. 2019 May 5;9(5):e025531. doi: 10.1136/bmjopen-2018-025531. PMID 31061026